CLINICAL TRIAL: NCT06567665
Title: Leucine Supplementation Strategies to Enhance Muscle Anabolic Responses in Older Age
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 23046
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Muscle Protein Synthesis
Keywords: Aging; Muscle protein synthesis; Leucine
MeSH Terms: interventions — Leucine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leucine supplementation between meals (Experimental): Volunteers will take leucine supplements between breakfast and lunch, between lunch and dinner, and between dinner and supper.
  Interventions: Dietary Supplement: Leucine
- Leucine supplementation with meals (Experimental): Volunteers will take leucine supplements with breakfast, with lunch and with dinner.
  Interventions: Dietary Supplement: Leucine

INTERVENTIONS:
Dietary Supplement: Leucine — Leucine is a dietary supplement that can be easily purchased over the counter at health food stores. It is an essential amino acid and is involved in stimulate muscle protein synthesis.

SUMMARY:
Sarcopenia describes the progressive decline of muscle mass and strength with advancing age and is associated with increased frailty and morbidity, however we do not currently have an effective treatment. Protein feeding and exercise is known to increase muscle mass, but aged muscle shows a lower response to these stimuli leading to muscle loss over time. We do know that ingesting leucine, a building block of protein, can overcome this reduced response to protein feeding and exercise leading to increased muscle mass in older people. However, we do not understand when the optimum time to ingest leucine is to maximise muscle mass after exercise in older people. In this study we will examine the effect of feeding leucine after exercise either with a meal or between meals.

ELIGIBILITY:
Inclusion Criteria:

* Male, 65-75 years of age
* BMI 18-28 kg/m2
* Non smoker
* Not performing regular resistance type exercise
* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* A BMI <18 or >28 kg·m-2
* Active cardiovascular disease: uncontrolled hypertension (BP > 160/100), angina, heart failure (class III/IV), arrhythmia, right to left cardiac shunt or recent cardiac event
* Cerebrovascular disease: previous stroke, aneurysm (large vessel or intracranial)
* Respiratory disease including pulmonary hypertension or chronic obstructive pulmonary disease (COPD)
* Metabolic disease: hyper and hypo parathyroidism, untreated hyper and hypothyroidism, Cushing's disease, types 1 or 2 diabetes (treated and untreated), inborn/ congenital errors of metabolism (e.g. phenylketonuria (PKU), galactosaemia)
* Active inflammatory bowel disease
* Acute infection
* Acute or chronic renal disease
* Malignancy (or history of malignancy with 5 y)
* Recent steroid treatment (within 6 mo), or hormone replacement therapy
* Coagulopathy
* Musculoskeletal or neurological disorders
* Known allergies to any of the product ingredients
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-08-05 (Estimated); Study Completion 2026-08-05 (Estimated)

PRIMARY OUTCOMES:
Muscle protein synthesis in response to leucine feeding | 7 days
  To quantify muscle protein synthesis in response to feeding leucine with a meal or in-between meals using mass spectrometry.

SECONDARY OUTCOMES:
Measure muscle anabolic and catabolic signalling pathways in response to leucine feeding | 7 days
  To determine the impacts of leucine feeding timings on muscle anabolic and catabolic signalling pathways using western blotting techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Brook, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell WK, Williams J, Atherton P, Larvin M, Lund J, Narici M. Sarcopenia, dynapenia, and the impact of advancing age on human skeletal muscle size and strength; a quantitative review. Front Physiol. 2012 Jul 11;3:260. doi: 10.3389/fphys.2012.00260. eCollection 2012. PMID 22934016
- [Background] Atherton PJ, Smith K. Muscle protein synthesis in response to nutrition and exercise. J Physiol. 2012 Mar 1;590(5):1049-57. doi: 10.1113/jphysiol.2011.225003. Epub 2012 Jan 30. PMID 22289911
- [Background] Wilkinson DJ, Bukhari SSI, Phillips BE, Limb MC, Cegielski J, Brook MS, Rankin D, Mitchell WK, Kobayashi H, Williams JP, Lund J, Greenhaff PL, Smith K, Atherton PJ. Effects of leucine-enriched essential amino acid and whey protein bolus dosing upon skeletal muscle protein synthesis at rest and after exercise in older women. Clin Nutr. 2018 Dec;37(6 Pt A):2011-2021. doi: 10.1016/j.clnu.2017.09.008. Epub 2017 Sep 23. PMID 29031484
- [Background] Katsanos CS, Kobayashi H, Sheffield-Moore M, Aarsland A, Wolfe RR. A high proportion of leucine is required for optimal stimulation of the rate of muscle protein synthesis by essential amino acids in the elderly. Am J Physiol Endocrinol Metab. 2006 Aug;291(2):E381-7. doi: 10.1152/ajpendo.00488.2005. Epub 2006 Feb 28. PMID 16507602
- [Background] Brook MS, Wilkinson DJ, Mitchell WK, Lund JN, Phillips BE, Szewczyk NJ, Greenhaff PL, Smith K, Atherton PJ. Synchronous deficits in cumulative muscle protein synthesis and ribosomal biogenesis underlie age-related anabolic resistance to exercise in humans. J Physiol. 2016 Dec 15;594(24):7399-7417. doi: 10.1113/JP272857. Epub 2016 Nov 7. PMID 27654940